CLINICAL TRIAL: NCT01494207
Title: Working on Wellness (WOW): A Worksite Health Promotion Intervention Programme
Brief Title: Working on Wellness (WOW) Intervention
Acronym: WOW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cape Town (Other)
Collaborators: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Tracy Kolbe-Alexander, Senior Lecturer, University of Cape Town
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: REC Ref 044/2009
Record Dates: First submitted 2011-12-14; First posted 2011-12-16 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-02

CONDITIONS: Physical Activity
Keywords: worksite; interventions; motivational interviewing; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle intervention (Experimental): Participants will receive the intervention (counseling) or usual care (control group)
  Interventions: Behavioral: Wellness counseling

INTERVENTIONS:
Behavioral: Wellness counseling — Each participant will receive up to six counseling sessions where the counselor will employ motivational interviewing techniques. The first and last session will be face-to-face with the remaining four sessions being telephonic.
  Other Names: Motivational Interviewing counseling

SUMMARY:
The main aim of this study is to measure the effectiveness of a worksite health promotion programme on improving physical activity behaviour and associated biological risk factors for cardiovascular disease among South African employees at increased risk for cardiovascular diseases. Additionally, the investigators will conduct an economic evaluation to determine the associated cost- effectiveness of these health related interventions offered at South African companies.

The investigators hypothesize that employees who receive the intervention counseling will have increased levels of physical activity and reduced risk for cardiovascular disease compared to those in the control group.

DETAILED DESCRIPTION:
Study Design:

"Working on Wellness - WOW" is a randomised controlled trial in South African worksites with a 12 month follow-up. Randomisation will take place at the company level, where participating companies will be assigned to either the intervention or the control group.

Study Population and Recruitment The study will be conducted in cooperation with a major national health insurer. Large companies (>300 employees) that are clients of this insurer, offering health and wellness days from August 2009 to February 2010 and that are based in Cape Town and Johannesburg will be approached to participate in this study.

Thereafter, over the course of two months all employees from these companies will be invited to participate in the wellness day(s) of their company. The invitation will take place as part of the feedback session at the wellness day and comprehensive information will be provided about the study. Employees agreeing to participate will be asked to sign an informed consent and to provide their email address and contact details. Participants will receive a small incentive at the start of the research study, and again upon completion.

Because all the companies hosting wellness days in this research study are clients of a major national health insurer, we will be able to access data for employees who do not volunteer for the screening activities. The data for the employees who choose not to participate will be sent to the researchers without any personal identifiers, thus ensuring employee confidentially. Being able to describe the non-responders is one of the strengths of this study design, and the insured population with whom we are working, providing insight into the problem of selection bias.

Control Group The employees in the control group will receive usual care. This comprises of feedback at the health and wellness day, referring employees to their physician if needed, and encouraging them to increase their level of physical activity and to improve nutrition in a generic way. They will receive general health promotion material detailing the risks for CVD and with advice on improving lifestyle behaviour. The participants from the control companies will also participate in follow up measurements at 6 and 12 months.

Intervention Group Individuals in the intervention group will receive the same advice and health promotion materials as those in the control group. Additionally, they will be offered an individually tailored intervention that consists of one-on-one counselling and educational materials. The counselling sessions will incorporate motivational interviewing techniques, to help the employee identify goals and strategies to improve their lifestyle.

An intervention mapping (IM) approach will be conducted at the start of the research study 13. This IM process will further inform the type and nature of intervention, including variables such as the optimal number of face-to face contacts and telephone contacts. Based on the research study by Groeneveld et al. it is envisaged that approximately two face to face and four telephone contacts will be required 8.

Outcome Measures

Health Risk Appraisal (HRA) Questionnaire The HRA is comprised of demographic, health and lifestyle factors, as well as questions related to stages of change for the various risk behaviours. The demographic variables include age and gender; while the lifestyle measures include smoking status, fruit and vegetable intake, habitual alcohol consumption and habitual physical activity. For smoking, fruit and vegetable intake and habitual physical activity, the participant also reports on readiness to change or improve these behaviours. The questions on readiness to change are based on the Transtheoretical Model stages of change 2.

Global Physical Activity Questionnaire Habitual physical activity will be measured using the 'Global Physical Activity Questionnaire' (GPAQ) 14. This is a self administered questionnaire that includes questions on habitual levels of light, moderate and vigorous activity. Furthermore, a sub sample of employees will be randomly selected to wear a pedometer for 4 consecutive days to measure the number of steps taken per day 15. This will provide a more objective measure of physical activity at baseline, 6 and 12 months.

Dietary Habits Habitual dietary fat intake will be measured using the Short Fat Questionnaire 16. In addition, participants will complete a food frequency questionnaire where they will record the type and amount of food consumed in an average week.

Presenteeism and Absenteeism The Healthy Days Questionnaire devised and tested by the US Centers for Disease control, will be used to measure health-related quality of life. Healthy days are calculated using a series of 4 questions, focusing on general perceived health, self-rated physical and mental health and the extent to which physical and/or mental health may have limited activity within the past 30 days 17. Absenteeism data will be obtained from the company's Human Resource office, in addition to the participant keeping a log book.

Clinical Measures All screening will conducted by qualified, trained staff, provided by the health insurer and will form part of their wellness day which is offered to their corporate clients. The following clinical measures will be performed at the wellness days.

Cholesterol screening will be conducted using finger-prick capillary blood samples (Accutrend ® GC analysers, Roche Diagnostics) to measure total serum cholesterol concentrations.

Blood pressure will be measured twice per person using an automated sphygmomanometer. Employees will be instructed to sit quietly for approximately three minutes before being measured.

Standing height (cm) will be measured to the nearest 0.1 cm, using a stadiometer. Body weight will be measured using a portable calibrated scale and recorded to the nearest 0.1 kg. Body Mass Index (BMI) will be calculated as body mass (kg) divided by height (m) squared (kg/m2).

Process Evaluation A process evaluation will be conducted to determine if the intervention was implemented as intended. The counselors and participants' will be required to critically appraise the various components of the intervention and to grade their experience. Fidelity intervention will be measured by the research team, using the MITI software to monitor contents and quality of interviews having taken place, attendance and number of missed and re-scheduled appointments).

Cost-effectiveness analysis The cost-effectiveness of the intervention programme will be determined from the societal perspective. The two main outcomes are the change in habitual physical activity levels and CVD risk profile to be determined by SCORE.

The intervention costs that will be included in models include the cost of the wellness days for NCD risk screening, training of counsellors, employment costs of counsellors, opportunity cost that may be lost if employee's sessions are during working hours, health promotion material, incentives, travel and telephone calls. Direct health care costs will be based on health-related claims data that will be obtained from the medical insurer. Indirect costs include costs for sickness absenteeism and costs for presenteeism. In addition, participants will keep a medical costs and absenteeism diary every 3 months.

Statistical Analyses STATISTICA software package was used for all the analyses (Stasoft, Inc. 184-199, Tulsa OK, SA) and intention to treat analysis will be performed for each of the outcomes. Mean, standard deviation and standard error will be calculated for the continuous variables. Frequency tables will be used to determine the percentage of individuals at risk, and also for the stages of change data. Chi squared analysis will be done to compare the percentage of employees meeting physical activity recommendations before and after the intervention. An Analysis of Variance (ANOVA) will be performed to determine whether there were significant changes in physical activity habits and nutrition in the intervention and control groups at 6 and 12 months. Logistic regression analyses will be completed, both before and after adjusting for confounders such as age.

For the economic evaluation, cost effective ratio's will be calculated by dividing the difference between the mean total costs of the intervention and usual care groups, by the difference in the means effects (such as change in physical activity). The confidence intervals of all the ratios will be determined using the bootstrapping technique. Furthermore, each of the cost effective ratios will be graphically presented on a cost effectiveness plane.

ELIGIBILITY:
Inclusion Criteria:

Employees identified to be at 'increased' or 'high' risk for CVD are eligible to take part in the research study. Risk status will be determined by using the (Euro) SCORE 12, together with their habitual physical activity levels, and Body Mass Index. SCORE incorporates age, total cholesterol, blood pressure and smoking status. This score ranks individuals according to their level of risk, ranging from very low to very high 10-year risk of fatal CVD (Appendix 1). Those with a risk of 5% or higher will be considered eligible.

Independent of the risk score, employees who are inactive (i.e., who do not comply with at least 30 minutes of moderate to vigorous activity on at least 5 days per week), or who smoke, and employees who are overweight (i.e., Body Mass Index ≥ 25 kg/m2) also will be eligible to take part in the study. Other inclusion criteria include being older than 18 years and having a contract with employer until end of 12-month measurement period

Exclusion Criteria:

* Employees will be excluded for the following reasons: pregnancy, diagnosis or treatment of cancer, any other disorder that makes physical activity impossible. Contract workers whose employ with the company will end before the 12 month follow up measurement, will also be excluded from the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2009-11; Primary Completion 2011-05 (Actual); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of a worksite intervention on physical activity behavior | 12 months
  The Global Physical Activity Questionnaire will be used for self reported levels of physical activity. Weekly time spent in moderate and vigorous activity will be reported.

SECONDARY OUTCOMES:
Risk for cardiovascular disease | 12 months
  The risk for cardiovascular disease will be based on blood pressure and cholesterol measurements, Body Mass Index, smoking status and dietary behavior

CONTACTS AND LOCATIONS:
Overall Officials: Tracy L Kolbe-Alexander, PhD, Principal Investigator — University of Cape Town
Locations (1):
- University of Cape Town, Cape Town, South Africa

REFERENCES:
- [Derived] Kolbe-Alexander TL, Proper KI, Lambert EV, van Wier MF, Pillay JD, Nossel C, Adonis L, Van Mechelen W. Working on wellness (WOW): a worksite health promotion intervention programme. BMC Public Health. 2012 May 24;12:372. doi: 10.1186/1471-2458-12-372. PMID 22625844